CLINICAL TRIAL: NCT06716216
Title: A Phase 3, Randomized, Open-Label Trial Comparing Efficacy and Safety of BGM0504 Versus Semaglutide Once Weekly As Add-on Therapy to Metformin And/or Sulfonylureas in Patients with Type 2 Diabetes
Brief Title: A Study of BGM0504 in Participants with Type 2 Diabetes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Collaborators: BrightGene New Bio-Medical Technology(Wuxi) Co.Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGM0504-Ⅲ -T2DM-02
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: 5 mg BGM0504 5 milligrams (mg) BGM0504 administered subcutaneously (SC) once a week. (Experimental): Drug: BGM0504 Administered SC
  Interventions: Drug: Drug: 5 mg BGM0504 Administered SC
- Experimental: 10 mg BGM0504 10 mg BGM0504 administered SC once a week. (Experimental): Drug: BGM0504 Administered SC
  Interventions: Drug: Drug:10 mg BGM0504 Administered SC
- Active Comparator: 1 mg Semaglutide 1 mg semaglutide administered SC once a week (Active Comparator): Drug: Semaglutide Administered SC
  Interventions: Drug: Drug: Semaglutide Administered SC

INTERVENTIONS:
Drug: Drug: 5 mg BGM0504 Administered SC — Experimental: 5 mg BGM0504 5 milligrams (mg) BGM0504 administered subcutaneously (SC) once a week.
  Arms: Experimental: 5 mg BGM0504 5 milligrams (mg) BGM0504 administered subcutaneously (SC) once a week.
Drug: Drug:10 mg BGM0504 Administered SC — Experimental: 10 mg BGM0504 10 mg BGM0504 administered SC once a week.
  Arms: Experimental: 10 mg BGM0504 10 mg BGM0504 administered SC once a week.
Drug: Drug: Semaglutide Administered SC — Active Comparator: 1 mg Semaglutide
  1 mg semaglutide administered SC once a week
  Arms: Active Comparator: 1 mg Semaglutide 1 mg semaglutide administered SC once a week

SUMMARY:
This trial is conducted in China. The aim of the trial is to evaluate the efficacy and safety of BGM0504 versus semaglutide as add-on to metformin and/or sulfonylureas in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* ■ Have been diagnosed with type 2 diabetes mellitus (T2DM);

  * Metformin is used in screening : 1) After used stable-dose metformin (≥1500 mg/day) or maximum tolerated (< 1500mg but≥1000mg daily) for 8 weeks before screening； 2)Metformin treatment dose <1500mg/day at Screening and have not reached the maximum tolerated dose ；3) Metformin combined with daily fixed-dose sulfonylureas (minimum therapeutic dose on the drug label) had been stable for ≥8 weeks when entering the induction period.
  * Have a BMI ≥23 kilograms per meter squared (kg/m²) at screening;
  * Be of stable weight (± 5%) for at least 3 months before screening;
  * Have HbA1c between ≥7.5% and ≤11.0%；

Exclusion Criteria:

* ■ Previous diagnosis of type 1 diabetes, special type diabetes;

  * There are malignant tumors within 5 years before screening, or patients are in latent of clinical malignant tumors (except patients with skin basal cell carcinoma and squamous cell carcinoma, cervical carcinoma in situ, prostate carcinoma in situ or papillary thyroid carcinoma who have no recurrence after surgery).
  * Have had chronic or acute pancreatitis any time prior to study entry;
  * Known allergic constitution (allergy to 3 or more kinds of food or drugs), or allergy to GLP-1 receptor agonists, or severe allergic diseases (asthma, urticaria, eczematous dermatitis, etc.) at screening;
  * Mentally incapacitated or speech-impaired;
  * Suspected or confirmed history of alcohol or drug abuse;
  * Pregnant or lactating woman;
  * The investigator considers that there are any other conditions that make it inappropriate to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-11-14 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Hemoglobin A1c (HbA1c) | Week 0 to Week 32
  Change from baseline in HbA1c after 32 weeks of treatment.

SECONDARY OUTCOMES:
Change From Baseline in Body Weight | Week 0 to Week 52
  Change from baseline in body weight after 52 weeks of treatment.
Change From Baseline in Hemoglobin A1c (HbA1c) | Week 0 to Week 52
  Change from baseline in HbA1c after 52weeks of treatment.
Percentage of Participants With HbA1c Target Value of <7% | Week 0 to Week 52
  Percentage of Participants With HbA1c Target Value of <7% after 52weeks of treatment.
Percentage of Participants With HbA1c Target Value of <5.7% | Week 0 to Week 52
  Percentage of Participants With HbA1c Target Value of <5.7%after 52weeks of treatment.
Change From Baseline in Fasting Serum Glucose | Week 0 to Week 52
  Change from baseline in FPG after 52 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China